CLINICAL TRIAL: NCT03591536
Title: Effects of Pentoxifylline on Reducing Acute Kidney Injury , Inflammation and Oxidative Stress After Cardiac Surgery
Brief Title: Effects of Pentoxifylline After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: nooshin dalili (Other)
Responsible Party: Sponsor-Investigator, nooshin dalili, Assistant Professor of SBMU, Shahid Beheshti University of Medical Sciences
Organization: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SBU13463
Record Dates: First submitted 2018-05-23; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Oxidative Stress; AKI; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Pentoxifylline

STUDY DESIGN:
Intervention Model Description: double blind randomized clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: only principle investigator knew the drug from placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pentoxifylline oral (Other): 50 adult patient underwent elective CABG intervention to be administered will be receiving main drug (pentoxifylline )oral 400 mg' every 8 hours from three days before surgery and on the day of surgery effect of intervention regarding antioxidant
  Interventions: Other: Pentoxifylline
- placebo (Placebo Comparator): 50 adult patient underwent elective CABG received oral placebo pill resembling completely to pentoxifylline 400 mg, every 8 hours from three days before surgery and on the day of surgery
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Pentoxifylline — 400 mg pentoxifylline oral tablet from 3 days before surgery and on the day of surgery
  Other Names: pentoxifylline tablets
  Arms: pentoxifylline oral
Other: Placebo — oral placebo tablets from 3 days before surgery and on the day of surgery
  Arms: placebo

SUMMARY:
Acute Kidney Injury (AKI) is a common and serious post operative complication and may occur in up to 50% of all patients undergoing cardiac surgery and is associated with 8% mortality rate compared with 0.9% in non-affected patients and remains a major factor for post surgery adverse outcomes. Early interventions to prevent postoperative AKI can help decreasing morbidity and mortality in these patients. Using cardiopulmonary bypass during cardiac surgery triggers systemic inflammatory response and recruits pro-inflammatory cytokines such as tumor necrosis factor, interleukin -10 (IL-10) and Interleukin-6 (IL-6) accompanying with production of free oxygen radicals which provokes oxidative stress in the milieu of ischemic reperfusion injury. Pentoxifylline as a non-specific phosphodiesterase inhibitor, can suppress the production of some factors of inflammatory response and oxidative stress, probably prevent post surgery AKI with these mechanisms.

DETAILED DESCRIPTION:
This is a double blind randomized multicenter clinical trial, enrolling 100 consecutive patients undergoing elective Coronary Artery Bypass Graft Surgery (CABG). Patients randomly and within concealment method divided into two groups, one to receive oral pentoxifylline 400 mg every 8 hours from three days before surgery and the other group received placebo. All the intubation , surgery and weaning protocols were the same.

ELIGIBILITY:
Inclusion Criteria:

* The elective CABG candidate

Exclusion Criteria:

* refusal to sign the consent,
* collagen vascular disease,
* use of immunosuppressive agents, corticosteroids (> 3 days), methylxanthines, diltiazem or sodium nitroprusside,
* angiography in the past 7 days,
* hemorrhagic diathesis and coagulopathy,
* uncontrolled diabetes mellitus
* sepsis
* renal failure (sCr > 2 mg/dl),
* hepatic failure (AST (Aspartate transaminase) or ALT(alanine transaminase) > 40 U/L)
* urinary tract infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
change of creatinine level before and after cardiac surgery | change of serum creatinine level 24 hours , 72 hours and 96 hours after cardiac surgery
  change of serum creatinine level post CABG between pentoxifylline and placebo arms

SECONDARY OUTCOMES:
Oxidative stress | before and 24 hours after end of cardiac surgery
  change of serum malondialdehyde (MDA) level as the inflammatory marker before and 24 hours after cardiac surgery
inflammatory status | before and 24 hours after end of cardiac surgery
  change of serum IL-6 , TNF( tumor necrosis factor) , IL-8 between two arms post cardiac surgery
measuring change of (BMI) weight in kilogram and height in centimeters ratio | before and after end of cardiopulmonary bypass pomp
  using weight and height ratio for calculating BMI

IPD SHARING:
Plan to Share IPD: No
no plan